CLINICAL TRIAL: NCT03505164
Title: The Role of suPAR in Doxorubicin Induced Cardiomyopathy in Breast Cancer Patients: Causative vs. Predictor
Brief Title: The Role of suPAR Biomarker in Blood Samples of Breast Cancer Patients During and Post Doxorubicin Chemotherapy: Causative vs. Predictor
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Tochukwu Okwuosa, Tochukwu M. Okwuosa, DO, FACC, Assistant Professor of Medicine and Cardiology, Director of Cardio-Onc Services, Principal Investigator in the suPAR pilot study., Rush University Medical Center
Other Study IDs: 16022426
Record Dates: First submitted 2017-08-31; First posted 2018-04-23 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Doxorubicin Adverse Reaction; Cardiomyopathies, Secondary; Breast Cancer
Keywords: Doxorubicin; suPAR; Cardiomyopathy; Heart Failure; Breast Cancer
MeSH Terms: conditions — Cardiomyopathies; Breast Neoplasms; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are put in a Centrifugation machine to separate the plasma. The plasma is then kept in -70 to -80 degrees Fahrenheit. Each sample will be studied for suPAR levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks to find a causative or predictive aspect of the suPAR biomarker for heart failure in breast cancer patients receiving Doxorubicin drug chemo regimen.

suPAR is a circulating protein which can be found in blood and/or urine and is associated with both kidney and heart disease.

* Hypothesis 1: Higher suPAR at baseline will predispose to Doxorubicin-induced cardiomyopathy or heart failure, observed by histology (under the microscope and other lab techniques) in mouse models, and tested using heart ultrasound techniques in humans.
* Hypothesis 2: suPAR is a marker of Doxorubicin-induced cardiomyopathy or heart failure after exposure to Doxorubicin, observed by histology (under the microscope and other lab techniques) in mouse models, and tested in humans.

The study will look at suPAR's association with three other biomarkers called troponin, B-Type Natriuretic Peptide (BNP) and C- Reactive Protein (CRP) that are also associated with heart disease.

In this study, the patient will have blood drawn as a routine part of the cancer treatment. That is prior to starting the cancer therapy, then after the first 2 and last 2 doxorubicin cycles (4 cycles altogether); as well as at 3, 6, & 12 months after doxorubicin treatment. (6 Visits in total) The patient will also have an echocardiogram (echo, heart ultrasound) at each of these time points. The first of the six study echos is considered part of the routine care.

DETAILED DESCRIPTION:
* Hypothesis 1: Higher suPAR at baseline will predispose to DOX-induced cardiomyopathy to be observed by histology in mouse models, and tested using LVEF (Left Ventricular Ejection Fraction) assessment, and surrogate cardiovascular outcome measures as described in humans.
* Hypothesis 2: suPAR is a marker of DOX-induced cardiomyopathy after exposure to DOX, to be observed by histology in mouse models, and tested using surrogate cardiovascular outcome measures as described in humans.

  1. Patients meeting outlined eligibility criteria are identified by breast cancer physicians working in the Rush Cancer Center. After eligibility is verified, patients are approached by the study coordinators or research fellow to discuss participation in the trial while patients were being seen by their provider within the cancer center and given the informed consent form for review. Patients are contacted approximately one week later to answer questions and plan for baseline visit if interested in enrolling.
  2. After signing the informed consent form, patients are officially enrolled. The research nurse, study coordinator, or research fellow will conduct research visits at each of the six study time points outlined in the protocol: pre-chemo, post-2 cycles of doxorubicin, post-4 cycles of doxorubicin, 3 months post-doxorubicin, 6 month post-doxorubicin and 12 months post-doxorubin
  3. Each study visit consists of collecting lab work via blood draw as detailed in the protocol as well as an echocardiogram performed with strain.
  4. Results from each test are collected, reviewed by the PI and documented in the patient's study binder.
  5. Preliminary human results have not been analyzed at this time as there is currently insufficient data collected.

In the laboratory approach of the study, the investigators aimed to establish the role of suPAR in DOX induced cardiomyopathy. The risk for DOX induced cardiomyopathy is known to increase with an increase of the accumulative dose. The investigators therefore used two doses of DOX. One group of mice received weekly injections of DOX at 3mg/kg bodyweight for 6 week (accumulative dose of 18mg/kg: DOX18) whereas another group received an accumulative dose of 25mg/kg bodyweight (DOX25: 5 weeks, at 5 mg/kg bodyweight). Blood samples were taken before the first injection, in the middle of treatment and at the end of treatment or at the day of sacrifice. The bodyweight of the animals was constantly monitored throughout the study.

At time of sacrifice, the heart weight and tibia length of the mice were quantified and cells were isolated to determine cellular levels of reactive oxygen species (ROS), contractility and Ca handling properties.

DOX induced cardiomyopathy can manifest years after treatment. Tissue samples from hearts of the DOX18 and DOX25 treatment group were obtained and quantitative PCR (Polymerase Chain Reaction amplification) of the ventricular tissue will help us determine the changes in protein expression and cellular signaling that underlie these DOX induced changes in cellular function.

Blood samples obtained from the DOX18 and DOX25 mice will be analyzed for their level of suPAR to determine changes in suPAR over the duration of treatment and potential correlations of [suPAR] with the degree of cardiac dysfunction.

The data collected will be analyzed using a descriptive analysis with means and standard deviations for continuous variables and percentages for categorical variables. A paired t-test comparing the pre-post difference will be used to compare the differences in the groups comparing pre to post measures of myocardial damage based on histology for mouse models, and LVEF (Left Ventricular Ejection Fraction) for human data. Analysis will be performed using SAS (statistical analysis software).

The expected results from the data collected in this study aim to both gain an understanding of and describe the relationship of various covariates to primary outcomes.

It is expected to have 50 participants by the study end date. There is a trained team working on the study, insuring quality of data gathering, recruitment and enrollment of patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 64 years
* Undergoing chemotherapy in the Rush cancer center with a plan for doxorubicin (Adriamycin®) chemotherapy.

Exclusion Criteria:

* Patients with metastatic breast cancer - complicated chemotherapy regimens, higher mortality risk
* HER2 (human epidermal growth factor receptor 2) positive breast cancer patients planned for trastuzumab therapy
* Patients with baseline cardiomyopathy (reduced LVEF: less than 50%)
* Patients with prior cardiovascular history of myocardial infarction (MI), angina, Congestive Heart Disease (CHD) death, coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI) including percutaneous transluminal coronary angioplasty (PTCA) and end-stage renal disease (ESRD), atrial fibrillation prior to cancer diagnosis
* Atrial fibrillation noted on baseline ECG

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients aged between 18 and 64, recently diagnosed with non metastatic breast cancer, and will be receiving doxorubicin containing chemo regimen.
  All patients are being treated at Rush University Medical Center, Chicago, IL, and Rush Oak Park Hospital, Oak Park, IL.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Causality relationship between the suPAR blood level and doxorubicin-induced cardiomyopathy | 12 months
  A blood draw will be done at baseline for all participants. The blood samples will be processed by Centrifugation, to separate the plasma, and the suPAR level measured using ELISA technique, to stratify the participants that have a higher or normal baseline.
  Although there is no current consensus regarding normal suPAR blood level, a level of 3000 pg/mL is considered a high level.
  Higher baseline blood level of suPAR, will predispose patients with breast cancer undergoing chemo regimen containing doxorubicin, to develop heart toxicity (heart failure or cardiomyopathy).
  Heart failure or Cardiomyopathy will be diagnosed by the clinical evaluation with signs and symptoms, LVEF (Left Ventricular Ejection Fraction) with echocardiograms (heart ultrasound), and surrogate cardiovascular outcome measures as described in humans, and tissue visualization and histology in mouse models, with various staining techniques, whether it was H&E staining, or other immunological staining.
Predictive relationship between suPAR blood level and doxorubicin-induced cardiomyopathy | 12 months
  A blood draw will be done at baseline for all participants. The blood samples will be processed by Centrifugation to separate the plasma, and the suPAR level measured using ELISA technique, to stratify the participants having a higher or normal baseline.
  Although there is no current consensus regarding normal suPAR blood level, a level less than 3000 pg/mL is considered a normal level.
  A normal baseline blood level of suPAR, with progressive elevation following doxorubicin exposure, along with other blood markers for heart failure, will be considered as a predictive marker for doxorubicin-induced cardiomyopathy.
  Heart failure or Cardiomyopathy will be diagnosed by the clinical evaluation with signs and symptoms, LVEF (Left Ventricular Ejection Fraction) with echocardiograms (heart ultrasound), and surrogate cardiovascular outcome measures as described in humans, and tissue visualization and histology in mouse models using H&E staining, or other immunological staining techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Tochi Okwuosa, DO, FACC, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Rush Oak Park Hospital, Oak Park, Illinois

IPD SHARING:
Plan to Share IPD: Undecided